CLINICAL TRIAL: NCT03090503
Title: Open Flexible-dose Randomized Study of the Effectiveness of Second Generation Antipsychotics in First Episode Psychosis Patients: A 3-year Follow-up
Brief Title: Effectiveness of Second Generation Antipsychotics in First Episode Psychosis Patients: 3-year Follow-up
Acronym: PAFIP3_3Y
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fundación Marques de Valdecilla (Other)
Collaborators: Centro de Investigación Biomédica en Red de Salud Mental (Network); Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Principal Investigator, Benedicto Crespo-Facorro, Associate Professor of Psychiatry, Fundación Marques de Valdecilla
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROAC2014_3Y; 2013-005399-16 (EudraCT Number); 14-0312 (Other: AEMPS)
Record Dates: First submitted 2017-03-14; First posted 2017-03-24 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-06

CONDITIONS: Schizophrenia; Psychotic Disorders; Psychosis
Keywords: Antipsychotic agents; Treatment; Effectiveness; Aripiprazole; Risperidone
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Aripiprazole; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aripiprazole (Active Comparator): Oral, dose range 10-30 mg/day, once or twice a day during study duration.
  Interventions: Drug: Aripiprazole
- Risperidone (Active Comparator): Oral, dose range 1-6 mg/day, once or twice a day during study duration.
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Aripiprazole — Initial dose: 10 mg.
  Other Names: Abilify
  Arms: Aripiprazole
Drug: Risperidone — Initial dose: 2 mg.
  Other Names: Risperdal
  Arms: Risperidone

SUMMARY:
This study compares the efficacy and effectiveness of two of the second-generation antipsychotics (SGAs) most used in our society in the treatment of schizophrenia (Aripiprazole and Risperidone) and the investigators do within an assistance program of early-stage psychosis individuals of the Community of Cantabria, clinical reference for the treatment of this disease in the Spanish Autonomous Community. Patients are included in a prospective naturalistic study, open flexible-doses and randomized into one of two possible patterns of treatment that includes the protocol.

DETAILED DESCRIPTION:
At present there is no evidence of which antipsychotic treatment would be the choice for treating the appearance of a non-affective psychotic disorder. There are a number of second-generation antipsychotic drugs that have proven effective in controlling positive symptoms of the disease but carry a number of variable side effects so there is no evidence on the treatment of choice in the market. Few studies try to assess the adhesion of a first episode of psychosis as prolonged treatment in time. Thus the development of experimental studies comparing the effectiveness of such treatments in clinical practice is of high interest for clinical psychiatrists.

Study setting and financial support: data for the present investigation are being obtained from an ongoing epidemiological and three-year longitudinal intervention program of first-episode psychosis (PAFIP) conducted at the outpatient clinic and the inpatient unit at the University Hospital Marqués de Valdecilla, Spain. Conforming to international standards for research ethics, this program was approved by the local institutional review board. Patients meeting inclusion criteria and their families provide written informed consent to be included in the PAFIP. The Mental Health Services of Cantabria provided funding for implementing the program. None pharmaceutical company supplied any financial support to it.

Study design: this is a flexible-dose study of two neuroleptics (Aripiprazole and Risperidone) assigned at aleatory ratio 1:1. Rapid titration schedule (5-day), until optimal dose is reached, is a rule used unless severe side effects occur. At the treating physician's discretion, the dose and type of antipsychotic medication could be changed based on clinical efficacy and the profile of side effects during the follow-up period. Antimuscarinic medication, Lormetazepam and Clonazepam are allowed for clinical reasons. No antimuscarinic agents are administered prophylactically. Antidepressants (Sertraline) and mood stabilizers (lithium) are permitted if clinically needed.

Clinical assessment: the severity scale of the Clinical Global Impression (CGI) scale, the Brief Psychiatric Rating Scale (BPRS), the Scale for the Assessment of Positive symptoms (SAPS) and the Scale for the Assessment of Negative symptoms (SANS) are used to evaluate symptomatology. To assess general adverse event experiences the Scale of the Udvalg for Kliniske Undersogelser (UKU), the Simpson-Angus Rating Scale (SARS) and the Barnes Akathisia Scale (BAS) are used. The same trained psychiatrist (BC-F) completed all clinical assessments.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing their first episode of psychosis (First Episode of Psychosis is defined as that psychopathological state in which for the first time and regardless of its duration, the patient has enough severe psychotic symptoms to allow a diagnosis of psychosis, having received no specific psychiatric treatment for him).
* Living in the catchment area (Cantabria).
* No prior treatment with antipsychotic medication or, if previously treated, a total life time of adequate antipsychotic treatment of less than 6 weeks.
* Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria for brief psychotic disorder, schizophreniform disorder, schizophrenia, or schizoaffective disorder.

Exclusion Criteria:

* Meeting DSM-IV criteria for drug dependence.
* Meeting DSM-IV criteria for mental retardation.
* Having a history of neurological disease or head injury with loss of consciousness.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-06 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of Aripiprazole and Risperidone at long term as measured by Percentage of discontinuation | 3 years
  Percentage of discontinuation of the initially assigned treatment: patients who completed the 3 year follow-up assessment and changed initial antipsychotic. Four reasons for the discontinuation are recorded: 1.- insufficient efficacy; 2.- marked side-effects; 3.- patient reported non-adherence and 4.- other causes. If more than one reason for discontinuation is present, the most important reason according to the above ranking is selected. Antipsychotic treatment data (doses, discontinuation and concomitant medications) are registered every 6 months. Insufficient efficacy is established at the treating physician's judgment only after at least three weeks of treatment.

SECONDARY OUTCOMES:
Change in general psychopathology measured by BPRS at long term | 3 years
  Measured by changes in total score of the Brief Psychiatric Rating Scale (BPRS).
Change in overall clinical status measured by CGI at long term | 3 years
  Measured by changes in total score of the Clinical Global Impression (CGI).
Change in negative symptoms measured by SANS at long term | 3 years
  Measured by changes in total score of the Scale for the Assessment of Negative Symptoms (SANS).
Change in positive symptoms measured by SAPS at long term | 3 years
  Measured by changes in total score of the Scale for the Assessment of Positive Symptoms (SAPS).
Emergence of adverse events by using the Scale of the Udvalg for Kliniske Undersogelser (UKU) | 3 years
  Measured by UKU. Those treatment-emergent adverse events that occurred at a rate of at least 10% in either treatment group are considered.
Emergence of akathisia by using the Barnes Akathisia Scale (BAS) | 3 years
  Measured by BAS. Treatment-emergent akathisia is assessed by both baseline-to-end changes and newly emergent categorical changes.
Emergence of extrapyramidal symptoms by using the Simpson-Angus Rating Scale (SARS) | 3 years
  Measured by SARS. Extrapyramidal symptoms is assessed by both baseline-to-end changes and newly emergent categorical changes.
Remission rate at long term | 3 years
  Remission is defined according to Andreasen et al. (2005) criteria covering BPRS and SANS scores: 1.- a score of mild or less (≤3) on six predefined BPRS symptom items: grandiosity, suspiciousness, unusual thought content, hallucinations, conceptual disorganization and mannerisms; and 2.- SANS items scores of ≤2 simultaneously in all items. These criteria are required to be maintained for at least 6 months.
Relapse rate at long term | 3 years
  Among patients who achieved clinical improvement and stability (CGI rating ≤ 4 and a decrease of at least 30% on BPRS total score and all BPRS key symptom items, by being rated ≤ 3 for more than 4 consecutive weeks at some point during the first 6 months following program entry), relapse is defined as any of the following criteria that occurred during follow-up: 1 - a rating of either 5 or above on any key BPRS symptom items, 2 - CGI rating of ≥ 6 and a change score of CGI of "much worse" or "very much worse", 3 - hospitalization for psychotic psychopathology, or 4 - completed suicide. The key BPRS symptoms are unusual thought content, hallucinations, suspiciousness, conceptual disorganization and bizarre behaviour. Exacerbation is defined as any 2-point increase of any of the key BPRS symptoms, excluding changes in which the rating remained at the non-psychotic level (i.e., <3).

CONTACTS AND LOCATIONS:
Overall Officials: Benedicto Crespo-Facorro, Professor, Principal Investigator — University Hospital Marqués de Valdecilla, IDIVAL, Department of Psychiatry, School of Medicine, University of Cantabria, CIBERSAM Centro Investigación Biomédica en Red Salud Mental, Santander, Spain.
Locations (1):
- University Hospital Marques de Valdecilla, Santander, Cantabria, Spain

IPD SHARING:
Plan to Share IPD: No